CLINICAL TRIAL: NCT03340493
Title: EXTEND-IA TNK: Extending the Time for Thrombolysis in Emergency Neurological Deficits - Intra-Arterial Using Intravenous Tenecteplase Part 2
Brief Title: Determining the Optimal Dose of Tenecteplase Before Endovascular Therapy for Ischaemic Stroke (EXTEND-IA TNK Part 2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neuroscience Trials Australia (Other)
Collaborators: The Florey Institute of Neuroscience and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTA1401a
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Pathologic Processes; Brain Infarction; Brain Ischemia; Tenecteplase; Fibrinolytic agents; Fibrin Modulating agents; Molecular Mechanisms of Pharmacological Action; Plasminogen; Tissue Plasminogen Activator
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia; Cerebral Infarction; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Pathologic Processes; Brain Infarction; Brain Ischemia | interventions — Tenecteplase

STUDY DESIGN:
Intervention Model Description: Patients will receive either intravenous tenecteplase (0.4mg/kg, maximum 40mg, administered as a bolus over ~10 seconds) or intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over ~10 seconds).
Who Masked: Outcomes Assessor
Masking Description: Blinded core laboratory adjudication of the primary outcome. NIHSS and mRS (secondary outcomes) performed by blinded assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Assigned Interventions (Active Comparator): Patients will receive intravenous tenecteplase (0.25mg/kg, maximum 25mg, administered as a bolus over ~10 seconds).
  Interventions: Drug: Tenecteplase
- Tenecteplase (Experimental): Patients will receive intravenous tenecteplase (0.4mg/kg, maximum 40mg, administered as a bolus over ~10 seconds).
  Interventions: Drug: Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — Tenecteplase 0.25mg/kg and 0.4mg/kg are being used
  Other Names: TNK

SUMMARY:
Patients presenting to the emergency department with acute ischemic stroke, who are eligible for standard intravenous thrombolysis within 4.5 hours of stroke onset will be assessed for major vessel occlusion to determine their eligibility for randomization into the trial. If the patient gives informed consent they will be randomised 50:50 using central computerised allocation to either 0.4mg/kg or 0.25mg/kg intravenous tenecteplase before all participants undergo endovascular thrombectomy. The trial is prospective, randomised, open-label, blinded endpoint (PROBE) design.

DETAILED DESCRIPTION:
The study will be a multicentre, prospective, randomized, open- label, blinded endpoint (PROBE), controlled phase 2 trial (2 arm with 1:1 randomization) in ischemic stroke patients.

Randomized patients will first be stratified by both the setting of treatment: metropolitan hospital vs regional hospital (>1 hour transfer to endovascular centre) vs mobile stroke unit; and by site of baseline arterial occlusion: Intracranial internal carotid artery (ICA) and Basilar artery versus Middle cerebral artery (MCA - M1 and M2); overall resulting in six strata.

Imaging is performed with CT or MR (magnetic resonance) acutely as part of standard care with imaging follow-up at 18-30 hours. The sequences and the parameters used follow the STIR (Stroke Imaging Research) roadmap guidelines, but imaging takes place acutely and at 18- 30hrs only, as previously validated.

The sample size estimation was based on the proportion of pre-endovascular reperfusion observed in the 0.25mg/kg group from Part 1 of EXTEND-IA TNK (22%). An estimated total sample size of 188 patients (with 94 patients in each of treatment and control arms) yielded 80% power to detect a significant difference of 20% in strata-weighted angiographic reperfusion (mTICI 2b/3) at initial angiogram (22% in 0.25mg/kg vs 42% in 0.4mg/kg arm) at two-sided statistical significance threshold of p=0.05 for superiority. Adaptive increase in sample size will be performed if the result of interim analysis using data from the first 150 patients is promising, as per the methodology of Mehta and Pocock.

During the trial, blinded analysis of operational characteristics revealed a 20% reduction in the time from thrombolysis to arterial access versus part 1 due to improved workflow (In the first 150 patients in part 2 median 37min [IQR 19-54] versus 46min [IQR 28-63] in part 1). This directly impacts the time for thrombolysis to have an effect. A 20% reduction in the hypothesized rate of reperfusion at initial angiogram (18% vs 33%) would require 145 patients per group. Allowing for potential further improvements in workflow the sample size re-estimation was postponed from 150 to 240 patients with a revised minimum sample of 300 patients. Adaptive increase in sample size will be performed if the result of interim analysis using data from the first 240 patients is promising, as per the methodology of Mehta and Pocock. The maximum sample size is capped at 656 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with acute ischemic stroke eligible using standard criteria to receive IV thrombolysis within 4.5 hours of stroke onset
* Patient's age is ≥18 years
* Arterial occlusion on CTA (computed tomography angiography) or MRA (Magnetic Resonance Angiography) of the ICA, M1, M2 or basilar artery.

Exclusion Criteria:

* Intracranial hemorrhage (ICH) identified by CT or MRI
* Rapidly improving symptoms at the discretion of the investigator
* Pre-stroke mRS score of ≥ 4 (indicating previous disability)
* Hypodensity in >1/3 MCA territory or equivalent proportion of basilar artery territory on non-contrast CT
* Contra indication to imaging with contrast agents
* Any terminal illness such that patient would not be expected to survive more than 1 year
* Any condition that, in the judgment of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
mTICI | Initial angiogram (day 0)
  Proportion of patients with substantial angiographic reperfusion (mTICI) score of 2b/3 (restoration of blood flow to >50% of the affected arterial territory) or absence of retrievable thrombus at initial angiogram.

SECONDARY OUTCOMES:
Modified Rankin Scale (mRS) | at 3 months post stroke
  mRS ordinal analysis. mRS 0-1 or no change from baseline and mRS 0-2 or no change from baseline.
National Institutes of Health Stroke Scale (NIHSS) | Initial angiogram (day 0)
  Proportion of patients with ≥8 point reduction in NIHSS or reaching 0-1 at 3 days (favourable clinical response) adjusted for baseline NIHSS and age
Symptomatic intracranial haemorrhage (SICH) | Within 36 hours post treatment
  SICH is defined as "Intracerebral hemorrhage (parenchymal hematoma type 2 - PH2 within 36 hours of treatment) combined with neurological deterioration leading to an increase of ≥4 points on the NIHSS"
Death | Up to 3 months post stroke
  Death due to any cause
Angiographic reperfusion | Up to 24 hours post treatment
  Proportion of patients with angiographic reperfusion adjusted for hyperdense clot length on non-contrast CT and time from thrombolysis to initial angiogram

CONTACTS AND LOCATIONS:
Locations (28):
- Australia (26):
  - Albury Hospital, Albury, New South Wales
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Brisbane, Queensland
  - Gold Coast University Hospital, Gold Coast, Queensland
  - Sunshine Coast University Hospital, Nambour, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Ballarat Health Services, Ballarat, Victoria
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Western Heath, St Albans, Victoria
  - Latrobe Regional Hospital, Traralgon, Victoria
  - North East Health Wangaratta, Wangaratta, Victoria
  - South West Healthcare, Warrnambool, Victoria
- New Zealand (2):
  - Auckland Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Yogendrakumar V, Beharry J, Churilov L, Pesavento L, Alidin K, Ugalde M, Weir L, Mitchell PJ, Kleinig TJ, Yassi N, Thijs VN, Wu TY, Brown H, Dewey HM, Wijeratne T, Yan B, Sharma GJ, Desmond P, Parsons MW, Donnan GA, Davis SM, Campbell BCV; EXTEND-IA TNK and Royal Melbourne Stroke Registry Investigators. Association of Time to Thrombolysis With Early Reperfusion After Alteplase and Tenecteplase in Patients With Large Vessel Occlusion. Neurology. 2024 Apr 9;102(7):e209166. doi: 10.1212/WNL.0000000000209166. Epub 2024 Mar 19. PMID 38502892
- [Derived] Yogendrakumar V, Churilov L, Mitchell PJ, Kleinig TJ, Yassi N, Thijs V, Wu T, Shah D, Bailey P, Dewey HM, Choi PMC, Ma A, Wijeratne T, Garcia-Esperon C, Cloud G, Chandra RV, Cordato DJ, Yan B, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM, Campbell BCV; EXTEND-IA TNK Investigators. Safety and Efficacy of Tenecteplase and Alteplase in Patients With Tandem Lesion Stroke: A Post Hoc Analysis of the EXTEND-IA TNK Trials. Neurology. 2023 May 2;100(18):e1900-e1911. doi: 10.1212/WNL.0000000000207138. Epub 2023 Mar 6. PMID 36878701
- [Derived] Sarraj A, Albers GW, Mitchell PJ, Hassan AE, Abraham MG, Blackburn S, Sharma G, Yassi N, Kleinig TJ, Shah DG, Wu TY, Hussain MS, Tekle WG, Gutierrez SO, Aghaebrahim AN, Haussen DC, Toth G, Pujara D, Budzik RF, Hicks W, Vora N, Edgell RC, Slavin S, Lechtenberg CG, Maali L, Qureshi A, Rosterman L, Abdulrazzak MA, AlMaghrabi T, Shaker F, Mir O, Arora A, Martin-Schild S, Sitton CW, Churilov L, Gupta R, Lansberg MG, Nogueira RG, Grotta JC, Donnan GA, Davis SM, Campbell BCV; SELECT, EXTEND-IA, EXTEND-IA TNK, and EXTEND-IA TNK Part-II Investigators. Thrombectomy Outcomes With General vs Nongeneral Anesthesia: A Pooled Patient-Level Analysis From the EXTEND-IA Trials and SELECT Study. Neurology. 2023 Jan 17;100(3):e336-e347. doi: 10.1212/WNL.0000000000201384. Epub 2022 Oct 26. PMID 36289001
- [Derived] Yogendrakumar V, Churilov L, Mitchell PJ, Kleinig TJ, Yassi N, Thijs V, Wu TY, Shah DG, Ng FC, Dewey HM, Wijeratne T, Yan B, Desmond PM, Parsons MW, Donnan GA, Davis SM, Campbell BCV; EXTEND-IA TNK Investigators. Safety and Efficacy of Tenecteplase in Older Patients With Large Vessel Occlusion: A Pooled Analysis of the EXTEND-IA TNK Trials. Neurology. 2022 Mar 22;98(12):e1292-e1301. doi: 10.1212/WNL.0000000000013302. Epub 2022 Jan 11. PMID 35017305
- [Derived] Ng FC, Churilov L, Yassi N, Kleinig TJ, Thijs V, Wu T, Shah D, Dewey H, Sharma G, Desmond P, Yan B, Parsons M, Donnan G, Davis S, Mitchell P, Campbell B. Prevalence and Significance of Impaired Microvascular Tissue Reperfusion Despite Macrovascular Angiographic Reperfusion (No-Reflow). Neurology. 2022 Feb 22;98(8):e790-e801. doi: 10.1212/WNL.0000000000013210. Epub 2021 Dec 14. PMID 34906976
- [Derived] Alemseged F, Ng FC, Williams C, Puetz V, Boulouis G, Kleinig TJ, Rocco A, Wu TY, Shah D, Arba F, Kaiser D, Di Giuliano F, Morotti A, Sallustio F, Dewey HM, Bailey P, O'Brien B, Sharma G, Bush S, Dowling R, Diomedi M, Churilov L, Yan B, Parsons MW, Davis SM, Mitchell PJ, Yassi N, Campbell BCV; BATMAN study group and EXTEND IA TNK study group. Tenecteplase vs Alteplase Before Endovascular Therapy in Basilar Artery Occlusion. Neurology. 2021 Mar 2;96(9):e1272-e1277. doi: 10.1212/WNL.0000000000011520. Epub 2021 Jan 6. PMID 33408145
- [Derived] Campbell BCV, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Dowling RJ, Yan B, Bush SJ, Thijs V, Scroop R, Simpson M, Brooks M, Asadi H, Wu TY, Shah DG, Wijeratne T, Zhao H, Alemseged F, Ng F, Bailey P, Rice H, de Villiers L, Dewey HM, Choi PMC, Brown H, Redmond K, Leggett D, Fink JN, Collecutt W, Kraemer T, Krause M, Cordato D, Field D, Ma H, O'Brien B, Clissold B, Miteff F, Clissold A, Cloud GC, Bolitho LE, Bonavia L, Bhattacharya A, Wright A, Mamun A, O'Rourke F, Worthington J, Wong AA, Levi CR, Bladin CF, Sharma G, Desmond PM, Parsons MW, Donnan GA, Davis SM; EXTEND-IA TNK Part 2 investigators. Effect of Intravenous Tenecteplase Dose on Cerebral Reperfusion Before Thrombectomy in Patients With Large Vessel Occlusion Ischemic Stroke: The EXTEND-IA TNK Part 2 Randomized Clinical Trial. JAMA. 2020 Apr 7;323(13):1257-1265. doi: 10.1001/jama.2020.1511. PMID 32078683
- [Derived] Campbell BC, Mitchell PJ, Churilov L, Yassi N, Kleinig TJ, Yan B, Thijs V, Desmond PM, Parsons MW, Donnan GA, Davis SM. Determining the optimal dose of tenecteplase before endovascular therapy for ischemic stroke (EXTEND-IA TNK Part 2): A multicenter, randomized, controlled study. Int J Stroke. 2020 Jul;15(5):567-572. doi: 10.1177/1747493019879652. Epub 2019 Sep 30. PMID 31564231